CLINICAL TRIAL: NCT01764178
Title: A Single Dose, Sequence-randomized, Open-label, 2x2 Crossover Study to Compare Pharmacokinetics Between Pitavastatn and Valsartan Co-administration and Livalo Complex Product in Healthy Male Subjects
Brief Title: To Evaluate the Safety and PK Characteristics in Healthy Volunteers-Livalozet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: JW-PTV-102A
Record Dates: First submitted 2013-01-01; First posted 2013-01-09 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2017-03

CONDITIONS: Hyperlipidemia; Hypertension
Keywords: Pitavastatin; Valsartan
MeSH Terms: conditions — Hyperlipidemias; Hypertension | interventions — pitavastatin; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Livalo fixed combination drug (Experimental): Livalo fixed combination drug(Pitavastatin + Valsartan)
  Interventions: Drug: Livalo fixed combination drug
- Pitavastatin + Valsartan (Active Comparator): Pitavastatin, Valsartan
  Interventions: Drug: Pitavastatin, Valsartan

INTERVENTIONS:
Drug: Livalo fixed combination drug — Pitavastatin 4mg / Valsartan 160mg
  Arms: Livalo fixed combination drug
Drug: Pitavastatin, Valsartan — Pitavastatin 4mg, Valsartan 160mg
  Other Names: Livalo, Diovan
  Arms: Pitavastatin + Valsartan

SUMMARY:
The purpose of this study is to compare pharmacokinetics between Pitavastatin and Valsartan co-administration and Livalo fixed combination drug in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Age 20-55 years at the time of Screening
* BMI 19-26 kg/m2 at the time of Screening

Exclusion Criteria:

* Received other investigational drug within 90 days prior to the first dose of study drug

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2013-01-22 (Actual); Primary Completion 2013-03-15 (Actual); Study Completion 2013-12-27 (Actual)

PRIMARY OUTCOMES:
Cmax and AUC of study drugs after single oral administration | 0-48hrs

SECONDARY OUTCOMES:
AUCinf of study drugs after single oral administration | 0-48hrs
t1/2β of study drugs after single oral administration | 0-48hrs
Tmax of study drugs after single oral administration | 0-48hrs

CONTACTS AND LOCATIONS:
Overall Officials: Kyun Seop Bae, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea